CLINICAL TRIAL: NCT02059850
Title: A Study to Determine the Feasibility of Treating Synovial Sarcoma and Myxoid/Round Cell Liposarcoma Using Autologous NY-ESO-1 Specific CD8+ T Cells With Cyclophosphamide Pre-conditioning But Without the Use of IL-2
Brief Title: NY-ESO-1 Specific T Cells After Cyclophosphamide in Treating Patients With Advanced Synovial Sarcoma or Myxoid/Round Cell Liposarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2720.00; NCI-2013-02464 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2720.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); K23CA175167 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Adult Synovial Sarcoma; Myxoid/Round Cell Liposarcoma; Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma, Synovial; Liposarcoma, Myxoid; Sarcoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cyclophosphamide, NY-ESO-1 specific T cells) (Experimental): Patients receive cyclophosphamide IV on days -3 and -2 and NY-ESO-1 specific T cells IV over 60 minutes on day 0. Patients may receive additional infusions at the discretion of the PI.
  Interventions: Biological: Autologous NY-ESO-1-specific CD8-positive T Lymphocytes; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Autologous NY-ESO-1-specific CD8-positive T Lymphocytes — Given IV
Drug: Cyclophosphamide — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best way to give NY-ESO-1 specific T cells after cyclophosphamide in treating patients with advanced synovial sarcoma or myxoid/round cell liposarcoma. Placing a gene that has been created in the laboratory into white blood cells may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving NY-ESO-1 specific T cells with cyclophosphamide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To confirm the safety and efficacy of cancer-testis antigen (NY-ESO-1) specific T cells (autologous NY-ESO-1-specific cluster of differentiation [CD]8-positive T lymphocytes) in patients with advanced synovial sarcoma and myxoid/round cell liposarcoma following conditioning with high dose cyclophosphamide.

SECONDARY OBJECTIVES:

I. To confirm the persistence of NY-ESO-1 tetramer positive cells in the peripheral blood at 10 weeks after T cell infusion for synovial sarcoma and myxoid/round cell liposarcoma patients receiving NY-ESO-1 specific T cells following cyclophosphamide conditioning but not post-infusion interleukin (IL)-2.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) on days -3 and -2 and NY-ESO-1 specific T cells IV over 60 minutes on day 0. Patients may receive additional infusions at the discretion of the Principal Investigator (PI).

After completion of study treatment, patients are followed up for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR SCREENING:

* Medical history including histopathological documentation of sarcoma
* Informed consent and Health Insurance Portability and Accountability Act (HIPAA) signing

CRITERIA FOR LEUKAPHERESIS:

* NY-ESO-1 expression in tumor by immunohistochemistry (IHC) is not required prior to screening consent; however, patients must have NY-ESO-1 expression to proceed with the leukapheresis; additionally patients must also meet the following criteria to proceed with leukapheresis (any exceptions to this will require prior approval by the Apheresis director and Principal Investigator):
* Physical exam and Karnofsky performance status
* Laboratory evaluation:
* Complete blood count (CBC), differential and platelet count
* Basic metabolic and hepatic function panels
* Puget Sound Blood Center Recipient Donor Battery Panel
* Pregnancy test for females of child-bearing potential
* Pulse > 45 and < 120
* Weight >= 45 kg
* Temperature =< 38 Celsius (C) (=< 100.4 Fahrenheit [F])
* White blood cell (WBC) >= 2,000
* Hematocrit (HCT) >= 30%
* Platelets >= 75,000
* Research blood including 40 mL of blood in a heparinized tube for peripheral blood mononuclear cell (PBMC) collection and 10 mL of blood for serum collection (generally in a red top tube) within 30 days of leukapheresis collection

INCLUSION CRITERIA FOR TREATMENT:

* A diagnosis of synovial sarcoma or myxoid/round cell liposarcoma
* Patients must have "advanced disease"; usually, this will mean metastatic disease; this may also be multiply recurrent disease or locally advanced disease; locally advanced disease is defined for this study as disease where a mutilating surgery is required and the patient is more likely than not to die of their disease despite an aggressive operation; patients with metastatic disease that has been resected or radiated are allowed to participate; Response Evaluation Criteria in Solid Tumors (RECIST) evaluable disease is not necessary for participation
* NY-ESO-1 positive by IHC (for this study, even a small level of positivity is acceptable); for patients with < 5% NY-ESO-1 by IHC positivity, the level of staining should be discussed with the patient and they should be informed that this will likely effect the efficacy of the therapy; this conversation must be documented in the patient's medical chart
* Human leukocyte antigen (HLA)-A0201 or HLA-A2402
* Zubrod performance status of '0-1'
* All patients must have an electrocardiogram (ECG) within 2 weeks of starting conditioning
* All patients must have a stress test within 6 months of starting treatment showing no evidence of cardiac ischemia
* All patients must have an echo or multi gated acquisition scan (MUGA) scan showing ejection fraction (EF) > 50% and normal troponin and creatine kinase (CK) myoglobin binding (MB) (echo may be done at the time of stress test as a stress echo); within 6 months of starting treatment; however if the patient has received cardiotoxic chemotherapy such as Adriamycin, they must have had an echo or MUGA scan since completing this treatment
* If there is a patient with an NY-ESO-1 expressing soft tissue sarcoma who would be otherwise eligible for the trial, which is either not synovial sarcoma (SS) or myxoid/round cell liposarcoma (MRCL) or there is controversy about the diagnosis, eligibility will be decided by the PI
* Patients must have NY-ESO-1 specific cells already produced or in production; these cells may be either in the process of their final expansion (for fresh infusion) or expanded and frozen at the time of enrollment

Exclusion Criteria:

* Patients for whom we are unable to generate NY-ESO-1 specific cells
* Pregnant women, nursing women, and men and women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative pregnancy test within two weeks prior to study entry
* Serum creatinine > 1.6 mg/dL or glomerular filtration rate < 50
* Serum glutamic oxaloacetic transaminase (SGOT) > 150 IU or > 3 x upper limit of normal
* Bilirubin > 1.6 mg/dL
* Prothrombin time > 1.5 x control
* Active symptomatic congestive heart failure
* Clinically significant hypotension (systolic blood pressure [SBP] < 80 mm HG or symptomatic)
* Newly diagnosed cardiac arrhythmia; patients with an arrhythmia that has been stable for at least 6 months will be allowed to participate
* Known untreated central nervous system (CNS) metastasis; patients with CNS metastasis will be allowed on study once treated
* Patients with active systemic infections requiring antibiotics or chronic maintenance/suppressive therapy; once the infection in question has resolved and patient is off antimicrobial treatment, patients may participate
* Systemic anticancer treatments (including chemotherapy and biologics) less than 3 weeks prior to T cell therapy; locally directed therapy (e.g. radiation) 2 weeks prior to cell infusion
* Known clinically significant autoimmune disorders requiring systemic immunosuppression for control
* Patients who are known to be human immunodeficiency virus (HIV) positive are not eligible for this study
* Current treatment with steroids
* Known infection with hepatitis B virus (HBV) and hepatitis C virus (HCV); (if a patient was not tested at the time of their leukapheresis, they must be tested prior to receiving T cell infusion; if testing was done for leukapheresis, this is adequate and does not need to be repeated)
* Patients with a known history of proven myocarditis, pericarditis, and/ or endocarditis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of grade III or greater toxicity graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | Up to 10 weeks
  The type and grade of toxicities noted during therapy will be summarized for each dose level. All adverse events noted by the investigator will be tabulated according to the affected body system. Descriptive statistics will be used to summarize changes from baseline in clinical laboratory parameters.

SECONDARY OUTCOMES:
Persistence of tetramer positive T cells | At 4 weeks
  The standard deviation and variance will be determined.
Persistence of tetramer positive T cells | At 10 weeks
  The standard deviation and variance will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States